CLINICAL TRIAL: NCT02836717
Title: Long Term Efficacy of Sacral Nerve Modulation (SNM) in Patients With Constipation or Stool Incontinence
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Lukas Marti, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: SGChir201601
Record Dates: First submitted 2016-06-22; First posted 2016-07-19 (Estimated); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-11

CONDITIONS: Constipation; Fecal Incontinence
Keywords: sacral nerve modulation; quality of life; stimulator maintenance; SNM
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: sacral nerve modulation — electric stimulation of the sacral nerve using an implanted electrode and stimulator

SUMMARY:
The aim of this study is to determine the success rate, the success duration, the complication rate, maintenance effort and quality of life several years after sacral nerve modulation (SNM) treatment for constipation or stool incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had received an SNM treatment in the last 10 years

Exclusion Criteria:

* pudendal nerve stimulation
* refusal to allow use of clinical data for retrospective data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients starting an SNM treatment for constipation or fecal incontinence between March 2006 and October 2015
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Marti, MD, Principal Investigator — Cantonal Hospital of St. Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Widmann B, Galata C, Warschkow R, Beutner U, Ogredici O, Hetzer FH, Schmied BM, Post S, Marti L. Success and Complication Rates After Sacral Neuromodulation for Fecal Incontinence and Constipation: A Single-center Follow-up Study. J Neurogastroenterol Motil. 2019 Jan 31;25(1):159-170. doi: 10.5056/jnm17106. PMID 30646487

RESULTS

PARTICIPANT FLOW:
Groups:
- FI Group: Patients suffering from fecal incontinence (only).
- Con Group: Patients suffering from fecal constipation (only).
- FI+Con Group: Patients suffering from fecal incontinence and constipation.
Period: Test Phase
Arm/Group | FI Group | Con Group | FI+Con Group
Started | 73 | 16 | 12
Completed | 59 | 8 | 12
Not Completed | 14 | 8 | 0
Not completed — Lack of Efficacy | 14 | 8 | 0
Period: Study Phase
Arm/Group | FI Group | Con Group | FI+Con Group
Started | 59 | 8 | 12
Completed | 45 | 1 | 11
Not Completed | 14 | 7 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lack of Efficacy | 8 | 6 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — abdominal surgeries | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FI Group | Con Group | FI+Con Group | Total
Number analyzed (Participants) | 73 | 16 | 12 | 101
Age, Continuous [Median (Full Range); unit: years] | 71 [25 to 87] | 72 [45 to 91] | 70 [34 to 89] | 72 [25 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 11 | 11 | 82
  Male | 13 | 5 | 1 | 19
Region of Enrollment [Number; unit: participants]
  Switzerland | 73 | 16 | 12 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Considering the Treatment a Success After 5 Years
Description: Treatment is considered a success if a patients reports a subjective 50% reduction in disease related complaints
Time Frame: 5 years
Population: Rate of successfully treated patients based on time-to-event ("Kaplan-Meier") statistic
Measure: Number (95% Confidence Interval); unit: percentage of success
Groups:
- All Patients: All patients in study
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
percentage of success | 81.7 [72.6 to 91.9] | 87.3 [78.1 to 97.6] | 31.2 [10.2 to 95.5] | 91.7 [77.3 to 100]

2. Secondary Outcome: Percentage of Patients Considering the Treatment a Success After 1 Years
Description: Treatment is considered a success if a patient reports a subjective 50% reduction in disease related complaints
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of success
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
percentage of success | 96.0 [91.7 to 100] | 98.2 [94.7 to 100] | 87.5 [67.3 to 100] | 91.7 [77.3 to 100]

3. Secondary Outcome: Percentage of Patients Considering the Treatment a Success After 3 Years
Description: Treatment is considered a success if a patient reports a subjective 50% reduction in disease related complaints
Time Frame: 3 year
Measure: Number (95% Confidence Interval); unit: percentage of success
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
percentage of success | 87.5 [80.2 to 95.5] | 90.3 [82.6 to 98.8] | 62.5 [36.5 to 100] | 91.7 [77.3 to 100]

4. Secondary Outcome: Number of Patients at Risk After 1 Year
Description: patients at risk according time-to-event statistics, i.e. number of participants still under evaluation, i.e. all participants minus the ones who have died, dropped out, or move out at the time of evaluation (https://en.wikipedia.org/wiki/Kaplan%E2%80%93Meier_estimator, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3059453/).
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
participants | 71 | 54 | 7 | 10

5. Secondary Outcome: Number of Patients at Risk After 3 Years
Description: as for outcome 4
Time Frame: 3 year
Measure: Number; unit: participants
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
participants | 53 | 39 | 5 | 9

6. Secondary Outcome: Number of Patients at Risk After 5 Years
Description: as for outcome 4
Time Frame: 5 year
Measure: Number; unit: participants
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 79 | 59 | 8 | 12
participants | 37 | 28 | 1 | 8

7. Secondary Outcome: Rate of Permanent Stimulator Implantations
Description: Rate of patients who finished the test phase with an external stimulator successfully (subjective reporting and 50% reduction of Wexner score for incontinence)
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients | FI Group | Con Group | FI+Con Group
Number analyzed (Participants) | 101 | 73 | 16 | 12
Participants | 79 | 59 | 8 | 12

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | FI Group | Con Group | FI+Con Group
All-Cause Mortality (participants affected / at risk) | 1/59 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 28/59 | 6/8 | 4/12
Other Adverse Events (participants affected / at risk) | 11/59 | 1/8 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FI Group (N=59) | Con Group (N=8) | FI+Con Group (N=12)
Other: Broken or dislocated lead (Product Issues) | 14 (19) | 3 (3) | 4 (5) — Stimulator lead broken or dislocated. Correct stimulation no longer possible
Device related infection (Infections and infestations) | 5 (6) | 1 (1) | 2 (2) — A disorder characterized by an infectious process involving the use of a medical device
Pain (General disorders) | 7 (8) | 2 (3) | 0 (0)
Other: Pulse generator dislocation (Product Issues) | 5 (5) | 0 (0) | 1 (1)
Other: Device failure (Product Issues) | 5 (5) | 1 (1) | 0 (0) — Loss of function of neural stimulator
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FI Group (N=59) | Con Group (N=8) | FI+Con Group (N=12)
Other: Dislocated lead (Product Issues) | 3 (3) | 0 (0) | 0 (0) — Stimulator lead dislocated. Correct stimulation no longer possible
Device related infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) — A disorder characterized by an infectious process involving the use of a medical device
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Other (Product Issues) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Observed death was unrelated to study treatment or study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes